CLINICAL TRIAL: NCT05856604
Title: Evaluation of Cognitive Effects Generated by Music Therapy for Older Adults With Cognitive Impairment Living in Care Homes - a Randomized Control Trial
Brief Title: Music Therapy for Older Adults With Cognitive Decline Living in Care Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Middlesex University (Other)
Collaborators: Methodist Homes for the Aged (Other)
Responsible Party: Principal Investigator, Anthony Mangiacotti, Principal Investigator, Middlesex University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ST020-2018
Record Dates: First submitted 2023-03-20; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Cognitive Impairment; Cognitive Decline
Keywords: music therapy; aging; cognitive rehabilitation; biomarkers; saliva cortisol/DHEA
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Experimental group = Improvisational Music Therapy Active control group = Storytelling activity
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Improvisational Music Therapy - 45min, one 2 one intervention.
  Interventions: Behavioral: Music Therapy
- Active Control (Active Comparator): Storytelling activity - 45min, one 2 one intervention.
  Interventions: Behavioral: Storytelling

INTERVENTIONS:
Behavioral: Music Therapy — Weekly individual (one2one) Music Therapy intervention lasting 4 months (n=16 sessions).
  Behavioral: Music Therapy Music therapy is a non-pharmacological intervention, in which music and its elements are used professionally as an intervention in medical, educational, and everyday environments with individuals, groups, families, or communities who seek to optimize their quality of life and improve their physical, social, communicative, emotional, intellectual, and spiritual health and wellbeing. This therapy has been shown to provide significant benefits for individuals with cognitive decline living in care homes, enhancing social-cognitive functions and reducing behavioural symptoms (Brotons & Koger, 2000; Hsu et al., 2015; Zhang et al., 2017).
  Arms: Experimental
Behavioral: Storytelling — Weekly individual (one2one) Storytelling intervention lasting 4 months (n=16 sessions).
  Behavioural: Storytelling is a non-pharmacological activity, in which a professional activity coordinator reads different stories (e.g., poems, novels) to the participants and used them to initiate a possible conversation.
  Arms: Active Control

SUMMARY:
This research aims to investigate whether the use of music-improvisation therapy for older adult participants can lead to improvements in cognitive ability levels, especially in attentional functions. Very relevant reviews highlight studies that demonstrate the effectiveness of Music Therapy training. However, only a few are based on randomised criteria and structured methodological approaches. This affects the generalizability of findings, as to whether Music Therapy interventions are effective in improving cognitive functions, mood, and quality of life of people with cognitive decline.

In order to make a difference, there is a need for more studies that are structured [i] according to rigorous empirical criteria (namely involving random assignment of participants to activity groups), [ii] and that gather scientific evidence, based on both standardized cognitive tests and biomarkers (hormones: Cortisol, or stress hormone, and DHEA or aging hormone; brain signal, EEG; Physiology: Respiratory Sinus Arrhythmia).

In this RCT study, the investigator investigated the effect of 4-month music therapy vs Storytelling program for older adults with cognitive decline, living in care homes.

DETAILED DESCRIPTION:
RESEARCH QUESTIONS

1. - What are the cognitive-neuropsychological benefits of Music Therapy activities in older adults with mild-moderate cognitive impairment?
2. - What are the behavioural-wellbeing benefits of Music Therapy activities in older adults with mild-moderate cognitive impairment?
3. - Can Music Therapy influence the psychophysiological domains (i.e., cortisol/DHEA ratio, RSA) of people with mild-moderate cognitive impairment?

Participants A power sample size calculation with an effect size (f) = 0.26, α= 0.05, Power (1-β) = 0.80 (any level over 0.80 is considered satisfactory) was performed with G*Power software yielding an overall n=32 minimum participant sample.

Participants were randomly allocated by a blind researcher to a MT (experimental group) or a ST intervention (active control group) using a computerised randomisation method.

To minimise a possible drop-out rate with a consequent loss of power, a total of 50 participants were recruited, of which 42 completed the study, 23 in the experimental group and 19 in the control group. All participants underwent a neuropsychological test battery examination. No baseline differences were found between the experimental and control group as to screening demographic variables, MMSE, Cognitive Reserve and a battery of cognitive and behavioural tests. Hence the two groups were equivalent at the start of the study.

DATA ANALYSIS Data of the neuropsychological, well-being and biomarker measures were analysed using a mixed design ANOVA with time (pre-post intervention) as a within-subject factor and group (MT vs ST) as a between-subjects factor. The dependent variables were the cognitive, neuropsychological test and biomarkers tests. Quantitative data were processed using IBM SPSS Statistic 25. Partial eta-square (ηp²) and Cohen's d were used as a measure of effect size.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥60yrs
* No significant hearing impairment that would negatively interfere with the music-based interventions
* Fluent in English
* Cognitive impairment: mild MMSE= 18-23, moderate MMSE= 10-17

Exclusion Criteria:

* Presence of severe motor deficits that would not allow individuals to participate in the intervention
* Having taken part in a cognitive training programme or Music Therapy programme within the last 6 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Music Cognitive Test (MCT) | Change in MCT score from baseline (time 0) to post-intervention period (+4 months).
  The Music Cognitive Test (Mangiacotti et al., 2022) which is a music-based cognitive screening test, specifically designed to measure possible changes brought by music-based interventions.
  The score range is 0-52 points; A higher score indicates better cognitive performance, with a score of 45 or above considered normal cognitive functioning.
Cornell Scale for Depression in Dementia (CSDD, Alexopoulos et al., 1988) | Change in CSDD score from baseline (time 0) to post-intervention period (+4 months).
  The Cornell Scale for Depression in Dementia (CSDD) is a test to screen depressive symptoms in older adults with dementia and cognitive impairment.
  Each item is rated for severity on a scale of 0-2 (0=absent, 1=mild or intermittent, 2=severe). The score range is 0-38 with scores above 10 indicating a probable major depression. Scores above 18 indicate a definite major depression.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA, Nasreddine et al., 2005) | Change in MoCa score from baseline (time 0) to post-intervention period (+4 months).
  The Montreal Cognitive Assessment (MoCA) is a brief extensively validated screening tool to measure cognitive impairment and is widely used in both clinical and experimental settings. The score range is 0-30 points; A higher score indicates better cognitive performance with a score of 26 or above considered normal cognitive functioning.
Verbal Fluency test, Phonemic & Semantic (VFT, Ardila et al., 2006; Machado et al., 2009) | Change in VTF score from baseline (time 0) to post-intervention period (+4 months).
  The Verbal Fluency test (VTF) is used to investigate lexical skills, semantic verbal fluency as well as the ability to organize an adequate research strategy. The total score for VFT is made by counting up the total number of animals (for the Semantic part) or words (for the Phonemic part) that the individual is able to produce. A higher score indicates better cognitive performance.
Clock Drawing test (CDT, Mondini et al., 2011) | Change in CDT score from baseline (time 0) to post-intervention period (+4 months).
  The Clock Drawing test (CDT) is used to evaluate praxis abilities, mental representation and planning abilities. The score range for CDT is 0-10 points with a higher score indicating better cognitive performance.
Tangled Figure Test (TFT, in Mondini et al., 2011, adaptation of Rey, 1964) | Change in TFT score from baseline (time 0) to post-intervention period (+4 months).
  The Tangle Figure Test (TFT) provides information on spatial-cognitive abilities and executive and naming difficulties. The score range for TFT is 0-50 with a higher score indicating better cognitive performance.
Trail Making Test (TMT-A, in Mondini et al., 2011) | Change in TMT-A score from baseline (time 0) to post-intervention period (+4 months).
  The Trail Making Test-A (TMT-A) assess selective attention and psychomotor speed. The test is scored based on how many seconds it takes the participant to complete the trial. Higher scores indicate a higher degree of cognitive impairment.
Bristol Activities of Daily Living Scale (BADL, Bucks et al., 1996) | Change in BADL score from baseline (time 0) to post-intervention period (+4 months).
  The Bristol Activities of Daily Living is a scale developed to measure activities of daily living (ADL) specifically designed for individuals with mild dementia living in a care home setting. The score range is 0-60, with a higher score indicating a higher degree of dependence on ADL.
Quality of Life in Alzheimer's Disease (QoL, Logsdon et al., 2002). | Change in QoL score from baseline (time 0) to post-intervention period (+4 months).
  The Quality of Life in Alzheimer's Disease (QoL) measures the quality of life in dementia. QoL is measured using the 13-item scale. Total score range from 13-52; higher scores indicate better quality of life.
The Satisfaction With Life Scale (SWLS, Diener et al., 1985). | Change in SWLS score from baseline (time 0) to post-intervention period (+4 months).
  The Satisfaction With Life Scale (SWLS) is a widely used 5-item measure of global life satisfaction and showed sufficient sensitivity to be a potentially valuable tool to detect changes in life satisfaction during clinical interventions (Pavot & Diener, 2009). The scale is a 7-point Likert-style response scale. The possible range of scores is 5-35 points.
Neuropsychiatric Inventory (NPI, Cummings et al., 1994) | Change in NPI score from baseline (time 0) to post-intervention period (+4 months).
  The Neuropsychiatric Inventory is a tool that provides information on behavioral symptoms commonly encountered in people with brain disorders. The total range score is 0-144 with a higher score indicating severe neuropsychiatric symptoms.

OTHER OUTCOMES:
Salivary Hormones index (cortisol/DHEA ratio) change from baseline/post (i.e., time 0/+4 months) | [Time Frame: Baseline vs. mid vs. post- intervention period (time 0/+2-months/+4months)
  Two types of salivary hormones will be collected: 1) Cortisol, which is associated with emotional distress and depressive symptoms (Herbert, 2013); 2) DHEA is an age-related hormone involved in different physiological mechanisms (anti-oxidant, anti-inflammatory; Kurata et al., 2004). The cortisol/DHEA ratio can be considered a reliable stress index (Theorell et al., 2021). The average of four daily collections will be performed to obtain a single daily value. Four passive-drool samples are collected in a single day for each participant:
  * At awakening (7am - 8am)
  * Before lunchtime (11.00am to 12.30am);
  * Before dinner (4pm to 5pm);
  * Evening (from 7pm to 8pm).
RSA change from baseline/post | Baseline and post- intervention period (time 0/+4 months)
  • Respiratory sinus arrhythmia (RSA): 5 min resting state based on Puyvelde et al., (2014)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Mangiacotti, PhD, Principal Investigator — Middlesex University
Locations (1):
- MHA Methodist Homes, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: No
the data have been analysed as group data (e.g., comparing men vs. women) and will be presented in an aggregate form

REFERENCES:
- [Background] Kim SJ, Yoo GE. Instrument Playing as a Cognitive Intervention Task for Older Adults: A Systematic Review and Meta-Analysis. Front Psychol. 2019 Feb 18;10:151. doi: 10.3389/fpsyg.2019.00151. eCollection 2019. PMID 30833913
- [Background] Fusar-Poli L, Bieleninik L, Brondino N, Chen XJ, Gold C. The effect of music therapy on cognitive functions in patients with dementia: a systematic review and meta-analysis. Aging Ment Health. 2018 Sep;22(9):1097-1106. doi: 10.1080/13607863.2017.1348474. Epub 2017 Jul 10. PMID 28691506
- [Background] Brotons M, Koger SM. The impact of music therapy on language functioning in dementia. J Music Ther. 2000 Fall;37(3):183-95. doi: 10.1093/jmt/37.3.183. PMID 10990596
- [Background] Hsu MH, Flowerdew R, Parker M, Fachner J, Odell-Miller H. Individual music therapy for managing neuropsychiatric symptoms for people with dementia and their carers: a cluster randomised controlled feasibility study. BMC Geriatr. 2015 Jul 18;15:84. doi: 10.1186/s12877-015-0082-4. PMID 26183582
- [Background] Zhang Y, Cai J, An L, Hui F, Ren T, Ma H, Zhao Q. Does music therapy enhance behavioral and cognitive function in elderly dementia patients? A systematic review and meta-analysis. Ageing Res Rev. 2017 May;35:1-11. doi: 10.1016/j.arr.2016.12.003. Epub 2016 Dec 23. PMID 28025173
- [Background] Mangiacotti, A., Cipriani, G., Ward, E., Franco, F., & Biasutti, M. (2022). Development and validation of the Music Cognitive Test: A music-based cognitive screening test. Psychology of Music, 030573562211008. https://doi.org/10.1177/03057356221100851
- [Background] Van Puyvelde M, Loots G, Vanfleteren P, Meys J, Simcock D, Pattyn N. Do you hear the same? Cardiorespiratory responses between mothers and infants during tonal and atonal music. PLoS One. 2014 Sep 10;9(9):e106920. doi: 10.1371/journal.pone.0106920. eCollection 2014. PMID 25207803
- [Background] Alexopoulos GS, Abrams RC, Young RC, Shamoian CA. Cornell Scale for Depression in Dementia. Biol Psychiatry. 1988 Feb 1;23(3):271-84. doi: 10.1016/0006-3223(88)90038-8. PMID 3337862
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Ardila, A., Ostrosky-Solís, F., & Bernal, B. (2006). Cognitive testing toward the future: The example of Semantic Verbal Fluency (ANIMALS). International Journal of Psychology, 41(5), 324-332. https://doi.org/10.1080/00207590500345542
- [Background] Machado TH, Fichman HC, Santos EL, Carvalho VA, Fialho PP, Koenig AM, Fernandes CS, Lourenco RA, Paradela EMP, Caramelli P. Normative data for healthy elderly on the phonemic verbal fluency task - FAS. Dement Neuropsychol. 2009 Jan-Mar;3(1):55-60. doi: 10.1590/S1980-57642009DN30100011. PMID 29213611
- [Background] ondini, S., Mapelli, D., Vestri, A., & Bisiacchi, P. S. (2011). Esame neuropsicologico breve 2: Una batteria di test per lo screening neuropsicologico. [A battery of tests for neuropsychological screening]. Raffaello Cortina Editore.
- [Background] Rey A (1958). L'examen clinique en psychologie (1st ed.). Paris: Presses universitaires de France
- [Background] Bucks RS, Ashworth DL, Wilcock GK, Siegfried K. Assessment of activities of daily living in dementia: development of the Bristol Activities of Daily Living Scale. Age Ageing. 1996 Mar;25(2):113-20. doi: 10.1093/ageing/25.2.113. PMID 8670538
- [Background] Logsdon RG, Gibbons LE, McCurry SM, Teri L. Assessing quality of life in older adults with cognitive impairment. Psychosom Med. 2002 May-Jun;64(3):510-9. doi: 10.1097/00006842-200205000-00016. PMID 12021425
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Pavot, W., & Diener, E. (2009). Review of the Satisfaction With Life Scale (pp. 101-117). https://doi.org/10.1007/978-90-481-2354-4_5
- [Background] Cummings JL, Mega M, Gray K, Rosenberg-Thompson S, Carusi DA, Gornbein J. The Neuropsychiatric Inventory: comprehensive assessment of psychopathology in dementia. Neurology. 1994 Dec;44(12):2308-14. doi: 10.1212/wnl.44.12.2308. PMID 7991117
- [Background] Herbert J. Cortisol and depression: three questions for psychiatry. Psychol Med. 2013 Mar;43(3):449-69. doi: 10.1017/S0033291712000955. Epub 2012 May 8. PMID 22564216
- [Background] Kurata K, Takebayashi M, Morinobu S, Yamawaki S. beta-estradiol, dehydroepiandrosterone, and dehydroepiandrosterone sulfate protect against N-methyl-D-aspartate-induced neurotoxicity in rat hippocampal neurons by different mechanisms. J Pharmacol Exp Ther. 2004 Oct;311(1):237-45. doi: 10.1124/jpet.104.067629. Epub 2004 Jun 2. PMID 15175425
- [Background] Theorell T, Engstrom G, Hallinder H, Lennartsson AK, Kowalski J, Emami A. The use of saliva steroids (cortisol and DHEA-s) as biomarkers of changing stress levels in people with dementia and their caregivers: A pilot study. Sci Prog. 2021 Apr-Jun;104(2):368504211019856. doi: 10.1177/00368504211019856. PMID 34030538
- [Derived] Mangiacotti AMA, Hsu MH, Barone C, Van Puyvelde M, Zandona A, Gabai G, Biasutti M, Franco F. Effects of one-to-one music therapy in older adults with cognitive impairment: A randomized controlled trial. Psychol Aging. 2024 Dec;39(8):960-982. doi: 10.1037/pag0000861. PMID 39666490
- See also: Aktas, A., & Keskin, B. (2013). Statistical power analysis. The 7th International Days of Statistics and Economics, 578-587 — http://msed.vse.cz/files/2013/224-Keskin-Burak-paper.pdf